CLINICAL TRIAL: NCT07138287
Title: Concerned Growth Factor Versus Miniral Trioide Aggregate in Management of Mature Permanent Molar of Children With Irreversible Pulpitis. An 18-month Randomized Control Trial
Brief Title: Concerned Growth Factor VS Miniral Trioide Aggregate in Treatment of Mature Permanent Teeth of Children With Symptomatic Irreversible Pulpitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Associate Professor of Pediatric and Community Dentistry, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3082
Record Dates: First submitted 2025-07-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Concerned Growth Factor Versus Miniral Trioide Aggregate in Management of Mature Permanent Molar With Irreversible Pulpitis
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Concerned Growth factor versus Miniral Trioide aggregate in management of Mature permanent Molar of children with irreversible pulpitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concerned Growth factor in management of Mature permanent Molar with irreversible pulpitis (Experimental)
  Interventions: Procedure: Concerned Growth factor in management of Mature permanent Molar with irreversible pulpitis

INTERVENTIONS:
Procedure: Concerned Growth factor in management of Mature permanent Molar with irreversible pulpitis — Concerned Growth factor in management of Mature permanent Molar of children with irreversible pulpitis
  Other Names: Pulpotomy

SUMMARY:
Concerned Growth factor versus Miniral Trioide aggregate in management of Mature permanent Molar of children with irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria: Permanent Molar with closed Apex and diagnosed with irreversible pulpitis

-

Exclusion Criteria:

* medically compromised children.

  * non restorable tooth
  * Necrotic tooth

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of cases using visual analogue scale, electrical pulp testing, Sensibility testing using both hot and cold and Percussion test for the teeth | 12 months
  Pain assessment using visual analogue scale pre operative, 6 hours post operative, 12hours post operative, 1 day post operative, 2 days post operative, 4 days, 1week, 2 weeks, 1month, 3 months, 6months and 1 year Sensibility test using thermal both hot and cold will be done pre operative and post operative Electrical pulp testing pre operative and post operative follow ups Percussion test to define any periapical or Periodontal issues
Radiographic evaluation of sucess of concentrated Growth factor versus Miniral Trioide aggregate in management of Mature permanent Molar with irreversible pulpitis | 12 months
  Standerdized periapical x rax will be performed before treatment, 3 months, 6minths, 9 months and one year after pulpotomy in the treated teeth to evaluated radiographic sucess

CONTACTS AND LOCATIONS:
Locations (1):
- Minya University Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We intend to share the data in BMC. We will share study protocol, materials and methods, results, discussion, recommendations and limitations of the current study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be available november 2025 and may ended at march 2026
Access Criteria: Any researcher who wants to have an access to my data can take it
URL: http://stda.minia.edu.eg/